CLINICAL TRIAL: NCT05240430
Title: Effectiveness of Mesenchymal Stem Cell in Patients With COVID-19 Associated SARS-CoV-2, Retrospective Clinical Study: When to Apply to Which Patient?
Brief Title: When to Apply to Which Patient in MSC?
Acronym: MSC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Trabzon Kanuni Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyfi KARTAL, MD, Assistant professor, Trabzon Kanuni Education and Research Hospital
Other Study IDs: Trabzon Kanuni TRH
Record Dates: First submitted 2022-01-27; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
Keywords: COVID-19; SARS-CoV-2; Mesenchymal Stem Cell; Intensive Care Units
MeSH Terms: conditions — COVID-19 | interventions — W8B2 protein, human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- stem cell application; Group I disease 0-7. days,: In mesenchymal stem cell application, according to the diagnosis of COVID 19 and the day of stem cell application; Group I disease 0-7. days,
  Interventions: Drug: Mesenchymal Stem Cell Antigen-1, Human
- stem cell application; Group II; 8-14 days of the disease. days: In mesenchymal stem cell application, according to the diagnosis of COVID 19 and the day of stem cell application; Group II; 8-14 days of the disease. days
  Interventions: Drug: Mesenchymal Stem Cell Antigen-1, Human
- stem cell application; Group III; those applied on the 15th day and after.: In mesenchymal stem cell application, according to the diagnosis of COVID 19 and the day of stem cell application; Group III; It will be divided into 3 groups as those applied on the 15th day and after.
  Interventions: Drug: Mesenchymal Stem Cell Antigen-1, Human

INTERVENTIONS:
Drug: Mesenchymal Stem Cell Antigen-1, Human — Human umbilical cord-derived MSCs were used in the study. MSCs were prepared/obtained/produced/provided by Atigen-Cell Technology Center, Trabzon, Turkey. MSC for patients was calculated as a single dose, 1x106 cells per kilogram. MSC was infused in 100 ml of normal saline at 2 ml/min over 40 min, as described in previous studies
  Other Names: Human umblical cord deriveted Mesenchymal Stem Cell

SUMMARY:
Mesenchymal stem cell (MSC) therapy is among the promising treatments for acute respiratory distress syndrome (ARDS). Our study aimed to investigate the clinical efficacy of MSC treatment in COVID-19 patients, to determine when this treatment can be applied to which patient, and to evaluate its contribution to prognosis.

DETAILED DESCRIPTION:
The study was conducted retrospectively in patients diagnosis of COVID-19 in the intensive care units. Patients with severe ARDS [partial pressure of arterial blood oxygen and inhaled oxygen fraction (PaO2: FiO2) ratio of 100 or less] were included in the study. Demographic data of the patients (gender, age), comorbidities (hypertension, coronary heart disease, diabetes, cerebrovascular diseases, hepatitis B infection, cancer, chronic kidney disease, and immunodeficiency), Charlson comorbidity index (CMI), date of diagnosis, date of admission to the hospital, date of admission to the ICU, Acute Physiology And Chronic Health Evaluation (APACHE) II score, presence of high flow nasal oxygen (HFNO) or mechanical ventilator (MV) support, laboratory findings (blood cell count, blood biochemistry, hepatorenal function, coagulation function, D-dimer, C-reactive protein (CRP), procalcitonin, ferritin, arterial blood gas analysis) before (day 0) and after MSC application, on 3rd and 7th days, partial oxygen/fractionated oxygen (Pa/Fi) ratio, discharge or death information, and attributed causes of death were recorded on the study form. Pa/Fi ratio was calculated with the formula (oxygen dissolved in arterial blood gas / oxygen liter given to the patient).

ELIGIBILITY:
Inclusion Criteria:

* Patients who were followed up and treated after being admitted to the Intensive Care Unit after March 2020
* Patients with COVID PCR +
* Typical or suspected cases of Thorax BT COVID
* Cases over the age of 18.

Exclusion Criteria:

* Those with a contraindicated condition (cancer disease, allergy) for MSC application
* Those who are endotracheal intubated during the application and are connected to a respirator
* Those who died in the first 24 hours after the application
* Cases that are not positive or suspicious for COVID.
* Cases under the age of 18.
* Cases where patient data could not be reached.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID PCR positive
  * Those who received MSC treatment
  * Those with advanced respiratory failure
  * Those who have progressed despite the standard recommended (antiviral, steroid, anticoagulant and vitamin) supportive treatment
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in acute phase reactants (C-reactive protein (CRP) after MSC administration in group I, II, III | MSC treatment Group I disease 0-7. days, Group II; 8-14 days of the disease. days, Group III; Those applied on the 15th day and after
  It was aimed to observe the changes in C-reactive protein (CRP), after MSC administration at different times (groups 1,2,3).
Change in acute phase reactants (procalcitonin) after MSC administration in group I, II, III | MSC treatment Group I disease 0-7. days, Group II; 8-14 days of the disease. days, Group III; Those applied on the 15th day and after
  It was aimed to observe the changes in procalcitonin after MSC administration at different times (groups 1,2,3).
Change in acute phase reactants ( white blood cell count) after MSC administration in group I, II, III | MSC treatment Group I disease 0-7. days, Group II; 8-14 days of the disease. days, Group III; Those applied on the 15th day and after
  It was aimed to observe the changes in white blood cell count after MSC administration at different times (groups 1,2,3).
Changes in respiratory support after MSC administration in Groups I, II, III | MSC treatment Group I disease 0-7. days, Group II; 8-14 days of the disease. days, Group III; Those applied on the 15th day and after
  It was aimed to observe the changes in respiratory support (such as high-flow nasal oxygen, mask with reservoir, and mechanical ventilation) after MSC administration at different times (groups 1,2,3).
Changes in arterial blood gas analysis (partial oxygen/fractionated oxygen (Pa/Fi) ratio) after MSC administration in Groups I, II, III | MSC treatment before (day 0) and after MSC application, on 3rd and 7th days,
  It was aimed to observe the changes in arterial blood gas analysis after MSC administration in Groups I, II, III.

SECONDARY OUTCOMES:
Effect on mortality after MSC administration in Groups I, II, III | 7, 14 and 28 days after MSC application
  The effect of MSC application at different times on mortality will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet AKYOL, MD, Study Chair — Trabzon Kanuni Training and Research Hospital, University of Healthy Sciences, Trabzon, Turkey
Locations (1):
- Trabzon Kanuni Training and Research Hospital, University of Healthy Sciences, Trabzon, Yomra, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No personal data belonging to the participants were used.

REFERENCES:
- See also: Mesenchymal stem cells derived from perinatal tissues for treatment of critically ill COVID-19-induced ARDS patients: a case series — https://pubmed.ncbi.nlm.nih.gov/33514427/
- See also: Treatment of severe COVID-19 with human umbilical cord mesenchymal stem cells — https://pubmed.ncbi.nlm.nih.gov/32811531/